CLINICAL TRIAL: NCT02749799
Title: An Open-Label, Multicenter Study of Patient-Reported Satisfaction Following Twice Daily Dosing With Betamethasone Dipropionate Spray, 0.05% in Subjects With Moderate Plaque Psoriasis
Brief Title: Patient Satisfaction Following Twice Daily Dosing With DFD-01 in Subjects With Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFD-01-CD-014
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — betamethasone-17,21-dipropionate; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DFD-01 (betamethasone dipropionate) Spray, 0.05% (Experimental): DFD-01 (betamethasone dipropionate) Spray, 0.05% to be applied twice daily on the affected areas (avoiding the face, scalp, groin, axillae and other intertriginous areas) for 28 days.
  Interventions: Drug: DFD-01 (betamethasone dipropionate) Spray, 0.05%

INTERVENTIONS:
Drug: DFD-01 (betamethasone dipropionate) Spray, 0.05% — DFD-01 (betamethasone dipropionate) Spray, 0.05% to be applied twice daily on the affected areas (avoiding the face, scalp, groin, axillae and other intertriginous areas) for 28 days.
  Other Names: Sernivo (betamethasone dipropionate, 0.05%) Spray

SUMMARY:
The purpose of this study is to assess clinical response and patient satisfaction when DFD-01 is used topically twice a day for moderate plaque psoriasis.

DETAILED DESCRIPTION:
This multicenter, multi-dose, open-label study was designed to assess clinical response and patient-reported satisfaction after dosing with DFD-01 twice daily for 28 days. The product was approved for the treatment of mild to moderate plaque psoriasis by the FDA on February 5, 2016 before the first patient was enrolled.

Forty five (45) adult males and females, 18 years of age and older with a clinical diagnosis of moderate plaque psoriasis who met inclusion/exclusion criteria were randomized at the Baseline Visit. Each site attempted to enroll 50% of the patients with 3% to 10% body surface area (BSA) involved and 50% of the patients with > 10% BSA involved.

The initial dose of study product was self-administered by the patient and supervised by clinic staff during the Baseline Visit. Patients continued to apply the study product to all affected areas (avoiding the face, scalp, groin, axillae or other intertriginous areas) twice daily (approximately 12 hours apart) for 28 days. Patients visited the clinic for a total of up to five scheduled visits:

* Screening (Day -60 to 1)*
* Baseline (Day 1)
* Interim Visit (Day 8 ± 2)
* Interim Visit (Day 14 ± 3)
* End of Study (Day 29 ± 3)

ELIGIBILITY:
Inclusion Criteria:

1. Patient understands the study procedures and agrees to participate by giving written informed consent. Patients must be willing to authorize use and disclosure of protected health information collected for the study.
2. Patient must be at least 18 years of age.
3. Patient must present with a clinical diagnosis of stable (at least 3 months) plaque-type psoriasis.
4. At least 3% Body Surface Area involved, not including the face, scalp, groin, axillae and other intertriginous areas.
5. Female patients of childbearing potential must agree to use contraception during the study which can include abstinence with an adequate secondary option should the patient become sexually active. A female is considered of childbearing potential unless she is:

   1. Postmenopausal for at least 12 months prior to study product administration;
   2. Without a uterus and/or both ovaries; or has been surgically sterile (i.e., tubal ligation) for at least 6 months prior to study product administration.

   Reliable methods of contraception are:
   1. Hormonal methods or intrauterine device in use > 90 days prior to study product administration; or
   2. Barrier methods plus spermicide in use at least 14 days prior to study product administration.
   3. Partner has had a vasectomy at least 3 months previous to study product administration.
   4. Essure® that has been in place for at least 3 months before the screening visit with radiograph confirmation of fallopian tube blockage.

   Exception: Sexually inactive female patients of childbearing potential are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided that they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study. An abstinent female must agree that if she becomes sexually active during the study she will use an acceptable form of contraception.

   All women must complete a urine pregnancy test at the Baseline Visit (Day 1) and the test result must be negative to be eligible for enrollment.
6. Patient must be in good general health as determined by the investigator and supported by the medical history and normal or not clinically significant abnormal vital signs (temperature, blood pressure and pulse).
7. Patient is physically able to apply study product to all affected areas or can obtain help.

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
2. Other inflammatory skin disease that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis).
3. Presence of pigmentation, extensive scarring, pigmented lesions, tattoos or sunburn that could interfere with the rating of efficacy parameters.
4. History of psoriasis unresponsive to topical treatments.
5. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
6. Ongoing infection (including viral lesions of the skin, fungal or bacterial skin infections, ulcers or wounds) or evidence of chronic infectious disease, history of or current system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation in the study.
7. Use within 180 days before Baseline Visit of biologic treatment for psoriasis (e.g., infliximab, adalimumab, etanercept, ustekinumab, secukinumab, or alefacept).
8. Have received treatment for any type of cancer within 5 years of the Baseline Visit, except skin cancer and cervical cancer (in situ) that are allowed if at least 1 year before the Baseline Visit.
9. Use within 60 days before the Baseline Visit of: 1) systemic or topical immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea) or 3) oral retinoids (e.g., acitretin, isotretinoin).
10. Use within 30 days before the Baseline Visit of: 1) systemic corticosteroids, 2) Ultraviolet light therapy, or 3) systemic anti-inflammatory agents* (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine). * Over-the-counter strength non-steroidal anti-inflammatory drugs used for transitional and common aches are permitted during the study.
11. Use within 14 days before the Baseline Visit of: 1) topical antipsoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene), 2) topical retinoids (e.g., tazarotene, tretinoin) or 3) topical corticosteroids.
12. History of unresolved or current hypothalamic-pituitary-adrenal suppression or significant endocrine disorder (Cushing's disease or Addison's disease) or uncontrolled diabetes.
13. Patients who have participated in a study of an investigational drug 30 days before the Baseline Visit.
14. Patients unable to comply with study requirements.
15. Female patients who are pregnant (or planning to become pregnant) or breast-feeding.
16. History of drug or alcohol abuse within the last year.
17. Planned use of a tanning bed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories Inc.
Locations (4):
- United States (4):
  - Site Four, Arlington Heights, Illinois
  - Site Two, New Albany, Indiana
  - Site One, Louisville, Kentucky
  - Site Three, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
Started | 45
Completed | 37
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 6
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
Percent Body Surface Area Involved [Mean (Standard Deviation); unit: Percentage of Body Surface Area] | 11.9 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Investigator's Global Assessment Grade
Description: The mean change in the IGA score from baseline to Day 14 was assessed. IGA score is a static assessment of disease severity and is based on overall severity of signs at each visit. It's a 4-point scale where '0' is absent disease and '4' is 'Severe/Very Severe' disease. A lower score at the end of the study compared to baseline (negative change), indicates an improvement in the disease condition.
Time Frame: Change from Baseline to Day 14.
Population: The ITT population included all randomized patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
Number analyzed (Participants) | 45
units on a scale | -0.8 (0.77)

2. Primary Outcome: Change in Percent Body Surface Area (BSA) Involved.
Description: Change in the BSA of involvement with psoriasis from baseline to Day 14 was assessed. BSA was assessed at Baseline, Days 8, 14 and 29.
Time Frame: Change from Baseline to Day 14.
Population: The ITT population included all patients randomized.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
Number analyzed (Participants) | 45
percentage of BSA | -1.3 (2.82)

3. Primary Outcome: Change in Dermatology Life Quality Index (DLQI)
Description: DLQI is a simple, compact, and practical questionnaire to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. The participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best. A lower score (i.e., negative change score) indicates improvement in the Quality of Life.
Time Frame: Change from Baseline to Day 14.
Population: The ITT population included all subjects randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
Number analyzed (Participants) | 45
units on a scale | -6.6 (6.72)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of informed consent up to the end of treatment (an average of 29 days).
Description: AEs were systematically recorded at every visit by direct questioning and in between the visits by the use of patient diaries. The patients could also call up the site staff directly by phone and report AEs. The AEs were recorded from the time of ICF signing up to the day of last treatment (an average of 29 days). The AEs were followed up until resolution, or lost to follow up, or death of the patient, or until 30 days after the last treatment administration.
Arm/Group | DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
All-Cause Mortality (participants affected / at risk) | 1/45
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-01 (Betamethasone Dipropionate) Spray, 0.05% (N=45)
Hip Fracture due to accidental fall (Injury, poisoning and procedural complications) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Acute kidney injury as a result of surgical complication following the hip fracture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No